CLINICAL TRIAL: NCT05132972
Title: Efficacy and Safety of Normoxic Allogenic Umbilical Cord Mesenchymal Stem Cells Administered as Adjuntive Treatment to Standard Treatment in Severe Patients With COVID-19
Brief Title: Allogenic UCMSCs as Adjuvant Therapy for Severe COVID-19 Patients
Acronym: UCMSC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia (Other Government)
Collaborators: Dr. Moewardi General Hospital, Surakarta, Indonesia (Other); Dr. Sardjito General Hospital, Yogyakarta, Indonesia (Unknown); Dr. Hasan Sadikin General Hospital, Bandung, Indonesia (Unknown); PT Bifarma Adiluhung (Industry)
Responsible Party: Principal Investigator, Bintang Soetjahjo, SpOT (K), MD. PhD, Coordinating Investigator, Dr. Moewardi General Hospital, Surakarta, Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRIN20211118a
Record Dates: First submitted 2021-11-23; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Covid 19
Keywords: COVID19; Mesenchymal Stem Cells (MCSs); Adjuvant therapy; Indonesia
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Group receiving standard COVID-19 treatment and UCMSC infusion
  Interventions: Biological: Normoxic Allogenic UCMSC
- Control (Sham Comparator): Group receiving standard COVID-19 treatment and normal saline infusion
  Interventions: Other: Normal saline solution

INTERVENTIONS:
Biological: Normoxic Allogenic UCMSC — Allogenic umbilical cord-derived mesenchymal stem cell (UCMSC) from normoxic, culture condition, administered through intravenousinfusion at dose 1x10^6 cells MSC/kg body weight. The treatment will be administered three times, at three days intervals (day 0, day 3, and day 6)
  Arms: Treatment
Other: Normal saline solution — Sterile saline solution and adminastered through intravenous infusion three times, at three day intervals (day 0, day 3, and day 6)
  Arms: Control

SUMMARY:
This study is conducted to assess the efficacy and safety of stem cells as adjunctive treatment for severe COVID-19 patients. Here, we want to study whether the administration of mesenchymal stem cells are safe and able to relieve some of the COVID-19 symptoms

DETAILED DESCRIPTION:
This is a randomized controlled trial. double-blind, multi-center clinical study conducted at three different hospitals, on 21 patients who received intervention and 21 patients who received control treatment. The purpose of this study is to evaluate the efficacy and safety of intravenous administration of normoxic allogeneic umbilical cord-derived mesenchymal stem cell (UCMSC) in the treatment group, compared to the control group who are only given standard COVID-19 treatments and normal saline infusion

ELIGIBILITY:
Inclusion Criteria:

* Man or woman age 18-75 years
* SARS-CoV2 positive as confirmed by SARS-CoV2 RT-PCR Test
* Diagnosed with pnumonia as confirmed by chect radiography and history of fever, coug with one of the following symptoms: RR > 30x per minute, SaO2 93%, FaO2/FiO2 300 mmHg
* Voluntarily joined the clinical trial and has signed the informed consent form

Exclusion Criteria:

* Pregnant and lactating woman
* Patient who are diagnosed or have history of tumor and cancer
* Patient whose mother or sister are diagnosed with breast or ovarian cancer
* Level of SGPT/ALT is ≥ 5 times upper limit from normal value
* Level of eGFR is < 30 ml/min
* Reluctant to sign informed consent and unwilling to take the required tests
* Require invasive ventilation
* Shock
* Organ failure
* Currently involve in other clinical trial, or join another clinical trial in the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-01-17 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Duration of hospital stay | 20 - 24 days
  Number of days since patient was administered until discharge in hospitals

SECONDARY OUTCOMES:
Post-administration clinical and radiological improvement | Baseline/day-1 (-2 days), day-15 (+/- 2 days), day-22 (+/1 2 days) post randomization day
  Chest X-ray evaluation; mMRC(Modified Medical Research Council) Dyspnea scale;
Adverse Event and Serious Adverse Event Evaluation | 20 - 24 days
  Evaluation of all adverse event or serious adverse event that is observed or reported by

CONTACTS AND LOCATIONS:
Overall Officials: Arief Nurudin, MD PhD, Principal Investigator — Dr. Moewardi General Hospital, Surakarta, Indonesia; Samekto Wibowo, Prof. MD, Principal Investigator — Dr. Sardjito General Hospital, Yogyakarta, Indonesia; Ahmad Faried, Prof. MD, Principal Investigator — Dr. Hasan Sadikin General Hospital, Bandung, Indonesia
Locations (3):
- Indonesia (3):
  - Dr. Moewardi General Hospital, Surakarta, Central Java
  - Dr. Hasan Sadikin, Bandung, West Java
  - Dr. Sardjito General Hospital, Yogyakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Atluri S, Manchikanti L, Hirsch JA. Expanded Umbilical Cord Mesenchymal Stem Cells (UC-MSCs) as a Therapeutic Strategy in Managing Critically Ill COVID-19 Patients: The Case for Compassionate Use. Pain Physician. 2020 Mar;23(2):E71-E83. PMID 32214286
- [Result] Richardson JB. Urban forests near municipal solid waste incinerators do not show elevated trace metal or rare earth element concentrations across three cities in the northeast USA. Environ Sci Pollut Res Int. 2020 Jun;27(17):21790-21803. doi: 10.1007/s11356-020-08439-3. Epub 2020 Apr 12. PMID 32281062
- [Result] Liang B, Chen J, Li T, Wu H, Yang W, Li Y, Li J, Yu C, Nie F, Ma Z, Yang M, Xiao M, Nie P, Gao Y, Qian C, Hu M. Clinical remission of a critically ill COVID-19 patient treated by human umbilical cord mesenchymal stem cells: A case report. Medicine (Baltimore). 2020 Jul 31;99(31):e21429. doi: 10.1097/MD.0000000000021429. PMID 32756149
- [Result] Galipeau J, Sensebe L. Mesenchymal Stromal Cells: Clinical Challenges and Therapeutic Opportunities. Cell Stem Cell. 2018 Jun 1;22(6):824-833. doi: 10.1016/j.stem.2018.05.004. PMID 29859173
- [Result] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Result] Khoury M, Cuenca J, Cruz FF, Figueroa FE, Rocco PRM, Weiss DJ. Current status of cell-based therapies for respiratory virus infections: applicability to COVID-19. Eur Respir J. 2020 Jun 4;55(6):2000858. doi: 10.1183/13993003.00858-2020. Print 2020 Jun. PMID 32265310